CLINICAL TRIAL: NCT06347562
Title: Next Generation Cytogenetics: Impact of New Technologies in the Genetic Diagnosis of Neurodevelopmental Disorders
Brief Title: Optical Genome Mapping for the Diagnosis of Neurodevelopmental Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 934
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Neurodevelopmental Disorder (Diagnosis)
MeSH Terms: conditions — Neurodevelopmental Disorders; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optical Genome Mapping (Experimental): explore the ability of Optical Genome Mapping (OGM) to detect known constitutional chromosomal aberrations.
  Interventions: Genetic: Optical Genome Mapping

INTERVENTIONS:
Genetic: Optical Genome Mapping — to evaluate the capability of OGM, its usefulness in clinical diagnosis, and its impact on genetic counseling.

SUMMARY:
to evaluate the ability of the Optical genome Mapping (OGM) approach to detect simple and complex constitutional chromosomal aberrations of clinical relevance, which had previously been identified with standard diagnostic approaches (karyotyping, FISH, CNV-microarray) in the context of neurodevelopmental disorders (NDDs) with/wo congenital anomalies (CA)

ELIGIBILITY:
Inclusion Criteria:

* subjects with neurodevelopmental disorders carrying a structural variant identified by standard cytogenetic analyses (Karyotyping/FISH/Chromosomal Microarray Analysis)

Exclusion Criteria:

* none

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-06-14 (Estimated); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Diagnostic concordance rate | 30 months
  percentage of concordance between optical genome mapping and standard assays (Karyotyping, Chromosomal Microarray Analysis) for all aberrations with clinical significance

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute E. Medea, Bosisio Parini, Lecco, Italy